CLINICAL TRIAL: NCT00309712
Title: Diabetes and Combined Lipid Therapy Regimen (DIACOR) Study: A Randomized, Double-Blind Study of Simvastatin, Fenofibrate, and Combined Fenofibrate and Simvastatin in Patients With Controlled Type II Diabetics Without Evidence of Coronary Disease
Brief Title: Diabetes and Combined Lipid Therapy Regimen (DIACOR) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Abbott (Industry); Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 128-009
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Type II Diabetes Mellitus; Mixed Dyslipidemia
Keywords: diabetes; combination lipid treatment; statin; fibrate; hypercholesteremia; mixed dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypercholesterolemia | interventions — Fenofibrate; Simvastatin

INTERVENTIONS:
Drug: fenofibrate 160 mg and placebo
Drug: simvastatin 20 mg and placebo
Drug: fenofibrate 160 mg and simvastatin 20 mg

SUMMARY:
The primary study hypothesis of this study is to determine whether there is a greater percentage of patients achieving a triglyceride level of <200 mg/dL with the combination of simvastatin 20 mg and fenofibrate 160mg than with either simvastatin 20 mg monotherapy or fenofibrate 160mg monotherapy.

DETAILED DESCRIPTION:
Diabetes is a strong risk factor for atherosclerosis and is often characterized by dyslipidemia with hypertriglyceridemia,low high-density lipoprotein (HDL), and modestly elevated low-density lipoprotein (LDL). Both HMG-CoA reductase inhibitors (statins) and fibrates improve lipoprotein metabolism and decrease coronary disease risk. Statins and fibrates affect different aspects of lipoprotein metabolism and each improve lipid metabolism complimentarily. Statins lower total cholesterol and LDL while fibrates decrease triglyceride concentrations and elevateHDL cholesterol. Since individual lipid parameters have been shown to be independent cardiovascular risk factors, it is especially important to target all lipid parameters to levels outlined in treatment guidelines.

The National Cholesterol Education Program Adult Treatment Panel ill (NCEP ill) guidelines have set target therapeutic levels for coronary heart disease (CHD) and CHD risk equivalents (including diabetes).Many patients, however, are not able to achieve optimal levels with a single lipid-controlling agent.

This is particularly evident among diabetics, who often have multiple dyslipidemias and are less likely to achieve effective lipid control.

Several small clinical trials have demonstrated that fibrate and statin dual therapy combine the specific effects of the two drugs by significantlyreducing total and LDL cholesterol while increasing HDL cholesterol, though problems are associated. Previous studies, conducted mainly with a gemfibrozil/cerivastatin combination, showed an increased incidence of side effects (myopathy, hepatotoxicity) and high cost. This problem was again addressed in a small study of74 patients randomized to combined or alternate-day simvastatin and fenofibrate therapy. Surprisingly, in this study, no cases of myopathy were reported, even among patients receiving combined simvastatin and fenofibrate therapy.

The Lipids in Diabetes Study (LDSH Study) examined the fenofibrate and cerivastatin combination in a large-scale trial of 4,000 patients. This study was stopped early because study treatment included cerivastatin, which was withdrawn from the United States market in 2001. Consequently, the results' utility will be limited in the United States.

Additional studies evaluating lipid therapies capable of meeting more aggressive treatment guidelines outlined in NCEP ill, especially among diabetic patients, are required. We propose a twelve-month study of simvastatin, micronized fenofibrate, and combination therapy among patients with controlled Type 2 diabetes mellitus. The primary objectives ofthis study will be to assess the safety and efficacy of combined micronized fenofibrate and simvastatin therapy versus micronized fenofibrate or simvastatin monotherapy. Secondary objectives will include evaluation of combined micronized fenofibrate and simvastatin therapy versus micronized fenofibrate or simvastatin monotherapy on novel lipid parameters and serological markers associated with significantly increased cardiovascular risk. The benefits of the study will be numerous. First, we will be able to detennine the efficacy of each treatment arm in achieving the more aggressive lipid level targets outlined in NCEP ill. Second, this trial, unlike previous studies, will assess the safety and efficacy of each treatment arm specifically among diabetic patients. Third, the length of therapy will allow adequate, yet efficient, evaluation of the tertiary endpoints, which include novel risk factors not previously assessed with combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Controlled Type n Diabetes Mellitus (HbAlc <9%)
2. Baseline levels ofLDL-C >100 mg/dL
3. HDL-C <40 mg/dL
4. Triglycerides :::200mg/dL and :::500mg/dL
5. ALT and AST levels :::30%above the ULN with no active liver disease and CK :::50%above the ULN
6. Alcohol consumption <2 drinks per day and with a maximum intake of <10 drinks per week
7. Patients who are currently treated with pioglitazone (15 to 45 fig/day), rosiglitazone (2 to 8 fig/day), or metformin (500 mg to 2500 fig/day) as monotherapy or in combination with insulin or sulfonylureas must have been on a stable dose of these anti-diabetic agents for the previous 3 months
8. Patients on warfarin or warfarin-like anticoagulants must agree to have their INRJPT levels drawn per standard of care by the local lab for adjustment of anticoagulant dosage

j. The patient understands the requirements of the study, and voluntarily agrees to participate in the study and provides informed consent

Exclusion Criteria:

1. Uncontrolled Type n Diabetes Mellitus (HbAlc >9%);
2. Known history of CAD
3. Known history of myopathy or rhabdomyolysis
4. Known history of intolerance to statins or fibric acid derivatives
5. The use of lipid lowering agents or treatments therapy including bile acid sequestrants, HMG-Co-A reductase inhibitors, fish oil, nicotinic acid (doses >200 mg/day) or niacin taken within 6 weeks prior to the eligibility for randomization visit or 8 weeks prior to the eligibility visit, if the patient is on fibrates
6. Serum creatinine> 1.5 mg/elL. If serum creatinine is between 1.2 and 1.49 mg/elL, the calculated creatinine clearance using the Crockcroft/Gault [Crockcroft, 1976 #124] formula must be >50 ml/min to be included in this study

Formula for Males:

CrCI= (140-age [years])x (body weight [kg]) (72) x (serum Cr [mg/elL])

Formula for Females:

CrCI=(140-age [years]) x (body weight [kg]) x 0.85 (72) x (serum Cr [mg/dL]) g. Active liver disease including viral hepatitis (hepatitis B or C) as determined by positive antibodies to core and surface antigen for hepatitis B, and positive antibodies for hepatitis C h. Uncontrolled hypertension (treated or untreated) with systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg i. Proteinuria as defined by >0.5 mg albumin per mg creatinine (if dipstick> 1+) or history of nephrotic syndrome j. Secondary hypercholesteremia due to hypothyroidism (TSH >6~U/mL) or nephrotic syndrome; Patients with a history of hypothyroidism, who are on a stable dose of thyroxine with normalized plasma thyroxine and TSH may be included k. Diagnosis of homozygous familial hypercholesteremia, or Types I or V hyperlipidemia 1. The concomitant use of cyclosporine; systemic itraconazole or ketoconazole, erythromycin or clarithromycin, nefazadone, or HIV protease inhibitors are excluded. The concomitant use of systemic (pO or IV) glucocorticoids, and verapamil (other calcium channel blockers are acceptable), or the consumption oflarge amounts of grapefruitjuice (> 1 quart) are excluded. m. Known hypersensitivity to any component of HMG-CoA reductase inhibitors or fibrates including history of elevated liver or muscle function tests, jaundice, or hepatotoxicity or myopathy associated with these treatments n. History of partial ileal bypass o. Treatment with any other investigational drug within the previous 30 days Currently using illicit drugs; history of drug or alcohol abuse within the past 5 years Type 1 diabetes mellitus, hyperlipidemicpancreatitis or known presence of cholelithiasis (gallstones); Any therapy or condition that would pose a risk to the patient or make it difficult for the patient to comply with requirements of the study s. Participation in any other studies involving investigational or marketed products within 30 prior to entryin the study. .

1. Pregnantand/orlactatingwomen,andwomenof childbearingpotentialnot usingacceptablemeansof contraception.Womenof childbearingpotentialmustbe usingadequatemeasuresof contraception(as determinedby the investigator)to avoidpregnancyandshouldbe highlyunlikelyto conceiveduringthe study period. Womenof childbearingpotentialmusthavea negativepregnancytest at the timeof initialscreening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-08; Study Completion 2006-09

PRIMARY OUTCOMES:
percent of patients achieving study goal oftriglycerides <200 mg/dL

SECONDARY OUTCOMES:
Percent of patients achieving all study goals: LDL-C < 100 mg/dL, HDL-C:40 mg/dL, Triglycerides <200 mg/dL and the Percent of patients achieving non-HDL cholesterol <130 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Muhlestein, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - McKay Dee Hospital, Ogden, Utah
  - LDS Hospital, Salt Lake City, Utah

REFERENCES:
- [Result] Muhlestein JB, May HT, Jensen JR, Horne BD, Lanman RB, Lavasani F, Wolfert RL, Pearson RR, Yannicelli HD, Anderson JL. The reduction of inflammatory biomarkers by statin, fibrate, and combination therapy among diabetic patients with mixed dyslipidemia: the DIACOR (Diabetes and Combined Lipid Therapy Regimen) study. J Am Coll Cardiol. 2006 Jul 18;48(2):396-401. doi: 10.1016/j.jacc.2006.05.009. Epub 2006 May 24. PMID 16843192